CLINICAL TRIAL: NCT02954471
Title: A Retrospective, Observational Molecular Epidemiology Study of HER2 Expression in Patients With Early / Metastatic Breast Cancer in Saudi Arabia
Brief Title: Study of Human Epidermal Growth Factor Receptor 2 (HER2) Expression in Participants With Early/Metastatic Breast Cancer in Saudi Arabia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29903
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Participants With Breast Cancer: This study will retrospectively collect data from participants with breast cancer in Saudi Arabia.

SUMMARY:
This is a retrospective, multicenter study, consisting of chart review of Saudi Arabian participants diagnosed with breast cancer between 2007 and 2013 and with available human epidermal growth factor receptor 2 (HER2) testing. Data on survival will be collected through 2015.

ELIGIBILITY:
Inclusion Criteria:

* Initially diagnosed with breast cancer
* Has a proven result of HER2 testing by immunohistochemistry (IHC), fluorescent in situ hybridization (FISH) or any other in situ hybridization (ISH) method
* Alive or not alive

Exclusion Criteria:

- Inconclusive, equivocal or unavailable result of HER2/neu overexpression by IHC and FISH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants With Early/Metastatic Breast Cancer in Saudi Arabia
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Positive HER2 Test Result | From January 2007 to December 2013 (Up to 7 years; assessed retrospectively)

SECONDARY OUTCOMES:
Percentage of Participants With Estrogen Receptor/Progesterone Receptor Positive Breast Cancer | From January 2007 to December 2013 (Up to 7 years; assessed retrospectively)
Percentage of Participants by Type of First-line and Subsequent Treatment Regimens Used | From January 2007 to December 2013 (Up to 7 years; assessed retrospectively)
Kaplan-Meier Estimate of Overall Survival (OS) | From January 2007 to December 2015 (Up to 9 years; assessed retrospectively)
Kaplan-Meier Estimates of Progression-free Survival (PFS) as Assessed Using Response Evaluation Criteria in Solid Tumors (RECIST) | From January 2007 to December 2013 (Up to 7 years; assessed retrospectively)
Percentage of Participants With Complete Response as Assessed Using RECIST | From January 2007 to December 2013 (Up to 7 years; assessed retrospectively)
Percentage of Participants With Partial Response as Assessed Using RECIST | From January 2007 to December 2013 (Up to 7 years; assessed retrospectively)
Percentage of Participants With Progressive Disease as Assessed Using RECIST | From January 2007 to December 2013 (Up to 7 years; assessed retrospectively)
Percentage of Participants with Stable Disease as Assessed Using RECIST | From January 2007 to December 2013 (Up to 7 years; assessed retrospectively)
Percentage of Participants With Adverse Events | From January 2007 to December 2013 (Up to 7 years; assessed retrospectively)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Saudi Arabia (3):
  - King Fahad Specialist Hospital; Oncology, Dammam
  - King Faisal Specialist Hospital & Research Centre, Jeddah
  - National Guard King Abdulaziz Medical City; Oncology, Riyadh